CLINICAL TRIAL: NCT03964675
Title: Evaluation of SenseGuard™ - a Noninvasive Respiratory Rate Measuring Device for Adult Patients
Brief Title: Evaluation of SenseGuard™- a Noninvasive Respiratory Rate Measuring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NanoVation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0137-18-NHR
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Condition
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory rate measurement (Experimental): Simultaneous measurement of respiratory rate using SenseGuard and Capnography
  Interventions: Device: SenseGuard

INTERVENTIONS:
Device: SenseGuard — A single invitational visit with a respiratory rate measurement duration of 30 minutes.

SUMMARY:
The SenseGuard™ is a new respiratory rate measuring and logging non-invasive device, and measures the respiratory rate by responding to changes in air moisture content in exhaled air. A prospective single-center, single arm study, designed to assess the bias, accuracy , precision and safety of the SenseGuard™ device in measuring of respiratory rate in adult patients. The study shall include a single invitational visit with a respiratory rate measurement duration of 30 minutes for each of 25 adult subjects hospitalized in internal wards.Subjects will be invited to participate should they meet all of the eligibility criteria. Following informed consent, subjects will be measured with both Microstream capnograph and SenseGuard™ measuring simultaneously so their results can be compared.

DETAILED DESCRIPTION:
Study description:

Respiratory rate (RR) is a vital sign used to monitor clinical condition of a patient. It is defined as the number of breaths per minute. Various devices using different techniques are available to measure RR. Currently this is measured at the bedside in clinical practice by counting the breaths, however the gold standard for measuring this vital sign is the capnograph. For the patient, this involves limiting the movement and talking so that the measurements can be taken.

A new respiratory rate measuring and logging device, SenseGuard™, is non-invasive and measures the respiratory rate by responding to changes in air moisture content (small amounts of water condensation) in exhaled air.

The study is planned as a prospective single-center, single arm study, designed to assess the bias, accuracy , precision and safety of the SenseGuard™ non-invasive device in measuring of respiratory rate in adult patients.

Subjects will be invited to participate should they meet all of the eligibility criteria. Following informed consent, subjects will be measured with both Microstream capnograph and SenseGuard™ measuring simultaneously so their results can be compared.

Study population:

25 hospitalized patients from Internal/General wards aged 18 and older.

Objective:

Evaluate the performance and safety of the SenseGuard™ non-invasive device in measuring respiratory rate in hospitalized adult patients.

Inclusion Criteria:

1. Hospitalized patients from the Internal/General wards.
2. Provision of signed and dated informed consent form
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Male or female, aged ≥18
5. Willing to adhere to the study regimen

Exclusion Criteria:

1. Intubated patients (i.e. endobronchial intubation) or patients currently undergoing a BPAP/CPAP treatment.
2. Presence of implanted electronic device intended to regulate cardiac activity (e.g., pacemaker or cardioverter/defibrillator)
3. Pregnancy or lactation
4. Known allergic reactions to materials used in the components of the SenseGuard™ system, i.e. polyethylene or silicon, or gold, nickel, copper or alloys containing any of the above.
5. Participation in another study in the last 4 weeks

Participant Duration:

A single invitational visit with a respiratory rate measurement duration of 30 minutes

Study Duration:

1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients from the Internal/General wards.
2. Provision of signed and dated informed consent form
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Male or female, aged ≥18
5. Willing to adhere to the study regimen

Exclusion Criteria:

1. Intubated patients (i.e. endobronchial intubation) or patients currently undergoing a BPAP/CPAP treatment.
2. Presence of implanted electronic device intended to regulate cardiac activity (e.g., pacemaker or cardioverter/defibrillator)
3. Pregnancy or lactation
4. Known allergic reactions to materials used in the components of the SenseGuard™ system, i.e. polyethylene or silicon, or gold, nickel, copper or alloys containing any of the above.
5. Participation in another study in the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of Respiratory Rate (RR) as measured by the SenseGuard™ system versus the gold standard (capnography). | 4 months
Frequency and incidence of any adverse events and serious adverse events related and unrelated to the device use | 4 months

SECONDARY OUTCOMES:
Usability (comfort and easiness) score of the SenseGuard™ system as measured by a questionnaire completed by the subjects | 4 months
  The easiness and comfort shall be evaluated using a questionnaire that includes 5 questions with possible scores ranging from 1(worst)-5(best)

CONTACTS AND LOCATIONS:
Locations (1):
- Galilee Medical Center, Nahariya, Israel